CLINICAL TRIAL: NCT03574285
Title: A Single-dose, Comparative Bioavailability Study of Two Formulations of Sarpogrelate HCl 300mg Tablets Under Feeding Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DDS17-035BE
Record Dates: First submitted 2018-06-20; First posted 2018-06-29 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anpl-one SR Tab. 300mg (Experimental): Anpl-one SR Tab. 300mg tablets followed by Sarpodipil SR Tab. 300mg tablets
  Interventions: Drug: Anpl-one SR Tab. 300mg; Drug: Sarpodipil SR Tab. 300mg
- Sarpodipil SR Tab. 300mg (Active Comparator): Sarpodipil SR Tab. 300mg tablets followed by Anpl-one SR Tab. 300mg tablets
  Interventions: Drug: Anpl-one SR Tab. 300mg; Drug: Sarpodipil SR Tab. 300mg

INTERVENTIONS:
Drug: Anpl-one SR Tab. 300mg — Anpl-one SR Tab. 300mg tablets followed by Sarpodipil SR Tab. 300mg tablets
  Other Names: Sarpogrelate HCl 300mg
Drug: Sarpodipil SR Tab. 300mg — Sarpodipil SR Tab. 300mg tablets followed by Anpl-one SR Tab. 300mg tablets
  Other Names: Sarpogrelate HCl 300mg

SUMMARY:
A Single-dose, Comparative Bioavailability Study of Two Formulations of Sarpogrelate HCl 300mg Tablets Under Feeding Conditions

DETAILED DESCRIPTION:
To evaluate the bioequivalence of two formulations of Sarpogrelate HCl 300mg, Anpl-one SR Tab. 300mg (Reference) and generic Sarpogrelate HCl 300mg (Test), after a single oral dose administration in healthy Thai volunteers under feeding condition: open label, single-dose, randomized, two-period, two-treatment, two-sequence, crossover, comparative bioavailability study

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking, male and female subjects, 19 years of age or older
* BMI ≥ 18.0 and ≤ 30.0 kg/m2.
* Females who participate in this study will be of childbearing or non-childbearing potential

Exclusion Criteria:

* Know history or presence of clinically significant neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, genitourinary, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the investigator, would jeopardized the safety of the subject or impact the validity of the study results

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration | 0-24hr
  Cmax
Area under the plasma concentration versus time curve | 0-24hr
  AUC

CONTACTS AND LOCATIONS:
Locations (1):
- Deawoong pharmaceutical, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No